CLINICAL TRIAL: NCT04146428
Title: Evaluating BOSCC and ELSA as Outcome Measures in the Context of a JASPER Intervention Trial
Acronym: EBJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Simons Foundation (Other)
Responsible Party: Principal Investigator, Connie Kasari, Ph.D., Professor/PhD, University of California, Los Angeles
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 19-001638
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder
Keywords: BOSCC; ELSA-T; JASPER; autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- clinician-mediated JASPER (Experimental): This group will consist of the child and therapist having one-on-one, JASPER sessions, twice a week.
  Interventions: Behavioral: clinician-mediated JASPER
- parent-mediated JASPER (Experimental): This group will consist of the therapist assisting the parent implement JASPER on the child twice a week.
  Interventions: Behavioral: parent-mediated JASPER

INTERVENTIONS:
Behavioral: clinician-mediated JASPER — JASPER is a developmentally anchored behavioral intervention that assumes that communication develops from social interactions in which specific social engagement strategies, symbolic representations, and early communication forms are modeled and naturally reinforced by the adult's responses to the child. The adult referred in this condition is the clinician/therapist.
  Arms: clinician-mediated JASPER
Behavioral: parent-mediated JASPER — JASPER is a developmentally anchored behavioral intervention that assumes that communication develops from social interactions in which specific social engagement strategies, symbolic representations, and early communication forms are modeled and naturally reinforced by the adult's responses to the child. The adult referred in this condition is the parent.
  Arms: parent-mediated JASPER

SUMMARY:
Research teams in Boston University, UCLA, and Weill Cornell will recruit 90 participants in 3 years (10 participants per site per year) and evaluate JASPER, play-based intervention, using the BOSCC and ELSA-T. Participants will be randomized to receive JASPER facilitated either by a clinician or the caregiver. After 10 weeks, the participants will be evaluated using the CGI to determine if they are "responders" or "non-responders". Nonresponders will be given a mix of clinician and caregiver-facilitated JASPER and responders will remain the course for the following 10 weeks. Coding of the BOSCC and ELSA-T will be the outcome measures and change will be evaluated throughout the study.

DETAILED DESCRIPTION:
Participants: 90 children with confirmed diagnoses of ASD (based on ADOS and clinical judgement) between 18 months and 5 years of age will be randomized into clinician-mediated vs. parent-mediated JASPER intervention at Weill Cornell (n=30; PI Dr. Kim), BU (n=30, PI Dr. Tager-Flusberg), and UCLA (n=30, PIs Drs. Lord & Kasari). Minimally verbal children eligible for the ADOS Toddler Module or Module 1 (pre or minimally verbal) or those who have emerging phrases who may receive Module 2 (phrase speech) will be enrolled. The sample will be limited to children with nonverbal mental ages greater than or equal to 12 months.

Pre-Intervention Behavioral Testing: We will administer the ADOS and Mullen Scales of Early Learning (MSEL), ESCS, SPA, and CCX. Parents will complete the interview version of the Vineland Adaptive Behavior Scales -3rd edition. In addition, the investigators will administer ELSA-T (following the same procedures that we developed in the first phase of this project described above) as well as the BOSCC with clinicians and caregivers (independent, standardized administration by caregivers). A subset of children (n=20) will be invited within a week of the first assessment for another ELSA/BOSCC sessions for test-retest reliability.

Responder vs. non-responder criteria: Children who show improvements in core ASD symptoms based on the treating therapists' CGI-Improvement ratings will be considered as "responders." Children who show stability or worsening on the CGI-I will be considered as "non-responders." Children will be stratified based on age and language levels across sites, and randomized into 10-week clinician- vs. caregiver- mediated JASPER interventions initially by the statistician at BU who will not be directly involved in the data collection. Both "responders" and "non-responders" will have monthly check-ins (2 total) with the research staff for an additional 10 weeks. Both groups will proceed to T3 assessments following the 20 weeks of treatment and check-ins.

At T2 (after first 10 weeks) and T3 (after 20 weeks, end of study), the investigators will again administer ELSA-T, BOSCC, as well as CGI, ESCS, SPA, and CCX.

Coding ELSA: Naïve coders will be trained to use ELAN to mark the beginning and end of each child speech vocalization/utterance and each examiner/parent utterance, which are coded on separate tiers. Coders will be blind about which kind of intervention the child received and when the ELSA recording was collected pre- or post-intervention. ELAN provides as output frequency of child utterances and frequency of adult utterances (corrected per unit time). The investigators have developed an algorithm that takes ELAN exported files containing the start and end time of each utterance from each speaker to derive a measure of conversation turn-taking (number of consecutive utterances produced by same speaker).

Note that these two measures are not independent, but clinical trials could define either one as a primary outcome measure depending on whether the targeted outcome focuses on the child's communicative abilities or social engagement. ELSA-T recordings will be collected at three sites, but all ELSA coding will be completed at BU.

Coding BOSCC: PI Dr. Kim's research team has trained, blind coders who will score the BOSCC without previous knowledge of the child and the time points of interactions. Different coders will be assigned for the clinician vs. caregiver BOSCC videos and for the parent behavioral coding. BOSCC videos will be collected at three sites, but all BOSCC coding will be done at Weill Cornell.

The same research activities will be conducted at UCLA, Boston University, and Weill Cornell.

ELIGIBILITY:
Inclusion Criteria:

* Minimally verbal children eligible for the ADOS Toddler Module or Module 1 (pre or minimally verbal) or those who have emerging phrases who may receive Module 2 (phrase speech) will be enrolled. The sample will be limited to children with confirmed diagnosis and nonverbal mental ages greater than or equal to 12 months. The child must be 18 months and 5 years of age.

Exclusion Criteria:

* Children that do not have a mental age greater than or equal to 12 months, don't have a confirmed diagnosis, are under the age of 18 months and older than 5 years of age.

Ages: 18 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-10-28 (Actual)

PRIMARY OUTCOMES:
Change in frequency of language utterances and number of conversation turns using the Elicitation of Language Samples for Analysis- Toddlers (ELSA-T) | Entry (1st month of the study), T2 (10 weeks after entry), T3 (20 weeks after entry)
  Dr. Tager-Flusberg's team created the ELSA, for collecting natural language samples (NLSs) from minimally to low verbal school-aged children and adolescents with ASD and developed a novel approach for deriving quantitative measures of linguistic communication (frequency of child utterances and number of conversational turns), in real-time from the language samples that could be useful for a range of clinical intervention trials. In this study, ELSA will be used on toddlers in this study, which has already been piloted.
Change in social communication using the Brief Observation of Social Communication Change (BOSCC) | Entry (1st month of the study), T2 (10 weeks after entry), T3 (20 weeks after entry)
  The BOSCC is a standardized measure of social communication change in children with ASD based on 12-minute videos of clinician- or caregiver-child interactions.

OTHER OUTCOMES:
ADOS Toddler Module or Module 1 or Module 2 (depends on child's language level) | Entry (1st month of the study)
  Confirm child's diagnosis.
Determine eligibility on nonverbal mental age using the Mullen Scales of Early Learning (MSEL) | Entry (1st month of the study)
  Nonverbal Development Quotients (DQ) (DQ; mental age ÷ chronological age)
Vineland Adaptive Behavior Scale- III | Entry (1st month of the study)
  The Vineland is a caregiver survey interview that measures the personal and social skills of individuals from birth through adulthood. The Adaptive Behavior Composite (ABC) scores range from 20 to 160 and indicate low (20-70), moderately low (70-85), adequate (85-115), moderately high (115-130), or high (130-160) overall adaptive functioning. Higher scores mean better outcome.
Demographic and Medical Questionnaire | Entry (1st month of the study)
  Descriptive measure to determine child's eligibility.No scores involved.
Presence of joint attention initiations using the Early Social-Communication Scales | Entry (1st month of the study), T2 (10 weeks after entry), T3 (20 weeks after entry)
  In this semi-structured interaction, the child and tester sit facing each other at a table with a set of toys in view but out of reach of the child which are introduced one by one (Mundy, Sigman, Ungerer, & Sherman, 1986; Seibert, Hogan, & Mundy, 1982). The joint attention initiations will then be coded.
Track the levels of spontaneous play acts using The Structured Play Assessment-R over the course of the study. | Entry (1st month of the study), T2 (10 weeks after entry), T3 (20 weeks after entry)
  SPA-R is designed to obtain the child's highest levels of spontaneous play acts. The child is presented with 5 different play sets by the experimenter; the entire play interaction last about 15-20 minutes. The child's play behaviors are videotaped and later coded. The variables of interest include the frequency of child initiated functional and symbolic play acts and also the count of different novel types of acts. This measure has shown excellent reliability and validity across a range of studies (Kasari et al., 2006; Sigman & Ruskin, 1999; Sigman & Ungerer, 1984).
Change in Joint Engagement on the Caregiver-Child Play Interaction (CCX) over the course of the study. | Entry (1st month of the study), T2 (10 weeks after entry), T3 (20 weeks after entry)
  A 10-minute interaction between parent and child. These sessions will be carried out with a standard set of toys and videotaped.
  Parents will be asked to engage their child in play as usual. Coders blind to child treatment assignment and time point will code the videotapes according to Adamson et al, 2004 coding procedures, the same as used in our previous studies (Harris, Kasari, & Sigman, 1996; Kasari et al, 2006; Kasari, et al, 2008). Joint engagement change will be recorded and measured throughout the study.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UCLA, Los Angeles, California
  - Semel Institute, Los Angeles, California
  - Boston University, Boston, Massachusetts
  - Weill Cornell Medical College/New York Presbyterian Hospital, White Plains, New York

IPD SHARING:
Plan to Share IPD: No
De-identified data will only be shared with researchers involved in the study.